CLINICAL TRIAL: NCT06337669
Title: Characterization of the Phenotypic Diversity in DupEx2 Duchenne Muscular Dystrophy and Identification of Predictive/Prognostic Markers
Brief Title: Characterization of DupEx2 Duchenne Muscular Dystrophy
Acronym: DMDDup2
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Previtali, Head Neuromuscular Repair Unit, IRCCS San Raffaele
Other Study IDs: OSRSCP-GUP21006
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for genomic analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To characterize the clinical phenotype and possible predictive/prognostic factors of patients with Duchenne muscular dystrophy (DMD) due to duplication of exon 2 (Dup2). Specifically, we aim 1) to describe the progression of motor, respiratory and cardiac function; 2) to enquire if the phenotypic spectrum of Dup2 is milder than classic DMD, 3) to perform whole genome sequencing (WGS) to characterize DNA breakpoints to correlate with the phenotype; 4) to collect material for future proteomic/transcriptomic studies.

Background/Rationale DMD is caused by mutations in the DMD gene and in 11% of cases is due to duplications. The most promising therapeutic approaches include mutation-specific therapies. Notably, there is increasing evidence that specific groups of mutations may underlie different disease trajectories compared to the "average" DMD population. It is thus mandatory to have more information on genotype-phenotype correlations and patterns of progression related to different genotypes.

Dup2 is the most common DMD duplication and the only one for which a AAV-mediated exon skipping study is ongoing. Despite most case series and databases ascribe Dup2 to severe phenotype, our preliminary findings sustain that these patients have collectively a milder progression of the disease and in 1/3 of cases a significantly milder phenotype. Moreover, our attempts to reveal mechanism involved in attenuating the phenotype would confute the hypothesis of alternative spicing transcripts as previously described for DMD with deletion of exon 2.

Research design and methods Clinical information regarding a cohort of 26 Italian Dup2 patients will be collected. Differences in time to loss of ambulation compared to a DMD control group will be achieved. Finally, we will retrieve DNA for correlative WGS studies.

Anticipated output We expect that Dup2 patients present a milder DMD phenotype , which might be predicted by genomic studies.

DETAILED DESCRIPTION:
The primary clinical endpoint is time to loss of ambulation (LOA).

Secondary endpoints include:

1. The change over time of the following functional measurements:

   1.1 Motor function: The 6 Minute Walk test (6MWT) and North Star Ambulatory Assessment (NSAA) including sub-items such as Time to Rise from the floor.

   1.2 Respiratory function: Forced Vital Capacity (FVC) Liters (L) and % of predicted; time to FVC% < 50%. Time to Nocturnal Ventilation initiation.

   1,3 Cardiac function: Left ventricular ejection fraction (EF) as measured by echocardiogram.
2. To characterize DNA breakpoints in mild vs severe phenotypes

ELIGIBILITY:
Inclusion Criteria:

* pediatric and adult DMD patients harboring a genetically confirmed duplication of the exon 2 in the dystrophin gene

Exclusion Criteria:

* patients lacking genetic confirmation of Dup2 mutation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Italian DMD patients with Dup2 mutation
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Age at loss of ambulation | 12 months
  Age at loss of ambulation

SECONDARY OUTCOMES:
Time test for motor function | 12 months
  The 6 Minute Walk test (6MWT) and North Star Ambulatory Assessment (NSAA) including sub-items such as Time to Rise from the floor.
Respiratory function | 12 months
  Forced Vital Capacity (FVC) Liters (L) and % of predicted; time to FVC% < 50%. Time to Nocturnal Ventilation initiation

CONTACTS AND LOCATIONS:
Overall Officials: Stefano C Previtali, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Dept. of Neurology, IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided